CLINICAL TRIAL: NCT07365410
Title: Furmonertinib 160mg Versus Furmonertinib 80mg Combined With Chemotherapy (Carboplatin + Pemetrexed) as First-Line Treatment for EGFR-Mutated NSCLC Patients With Brain Metastases: A Multicenter Study of Efficacy and Safety
Brief Title: Furmonertinib 160mg vs 80mg + Chemotherapy in EGFR-Mutated NSCLC With Brain Metastases: Efficacy and Safety Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20250722
Record Dates: First submitted 2025-11-26; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer (NSCLC); Brain Metastases; Furmonertinib; EGFR Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — aflutinib; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Furmonertinib 160mg Group (Experimental): Participants receive oral furmonertinib 160mg once daily as first-line treatment.
  Interventions: Drug: Furmonertinib
- Furmonertinib 80mg + Chemotherapy Group (Active Comparator): Participants receive oral furmonertinib 80mg once daily combined with intravenous carboplatin + pemetrexed (cycle-based) as first-line treatment.
  Interventions: Drug: Furmonertinib; Drug: carboplatin; Drug: pemetrexed

INTERVENTIONS:
Drug: Furmonertinib — Oral administration, 160mg once daily.
  Arms: Furmonertinib 160mg Group
Drug: Furmonertinib — Oral administration, 80mg once daily
  Arms: Furmonertinib 80mg + Chemotherapy Group
Drug: carboplatin — Intravenous infusion, cycle-based (per study protocol).
  Arms: Furmonertinib 80mg + Chemotherapy Group
Drug: pemetrexed — Intravenous infusion, cycle-based (per study protocol).
  Arms: Furmonertinib 80mg + Chemotherapy Group

SUMMARY:
This multicenter study evaluates the efficacy and safety of furmonertinib 160mg versus furmonertinib 80mg plus chemotherapy (carboplatin + pemetrexed) as first-line treatment for EGFR-mutated NSCLC patients with brain metastases. It aims to determine which approach is more effective and safer.

ELIGIBILITY:
IInclusion Criteria

* Aged 18 to 75 years (male or female)
* Histopathologically confirmed, unresectable, and non-radiocurable newly -diagnosed locally advanced or metastatic lung adenocarcinoma
* Confirmed by local laboratory to have one of the following EGFR mutations: -19Del or L858R (single or mixed mutations are allowed)
* Treatment-naive for locally advanced (not suitable for surgery/radiotherapy per investigator) or metastatic NSCLC; adjuvant/neoadjuvant therapy completed >6 months before first progression is allowed (≤6 months is considered pretreated)
* At least one measurable tumor lesion per RECIST 1.1 (lesions previously treated with radiotherapy are excluded; if only one measurable lesion exists, biopsy is allowed but baseline imaging must be performed ≥14 days after biopsy)
* Confirmed stable and asymptomatic brain metastases
* Sufficient organ function (per laboratory tests): ANC ≥1.5×10⁹/L, PLT ≥100×10⁹/L, HGB ≥90g/L; TBIL ≤1.5×ULN, AST/ALT ≤2.5×ULN (for liver metastasis: TBIL ≤3×ULN, AST/ALT ≤5×ULN); CrCL ≥50 ml/min (Cockcroft-Gault formula)
* ECOG performance status 0-2 (no significant disease deterioration in 2 weeks before screening)
* Expected survival >12 weeks after first dose
* Non-pregnant women of childbearing potential (no pregnancy plan); women and men agree to use effective contraception during the study and 6 months after drug discontinuation
* Voluntarily signs informed consent and understands the study procedures Exclusion Criteria（排除标准）
* NSCLC with predominantly squamous cell histology, small cell lung cancer, neuroendocrine carcinoma, or other non-adenocarcinoma histologies
* Concurrent positive for other driver genes (ALK fusion, ROS1 fusion, RET rearrangement, BRAF mutation, NTRK fusion, MET mutation, KRAS mutation); TP53, RB1, and BRAC mutations are excluded
* Expected to receive other anti-tumor therapies during the trial
* Major surgery (except vascular access or biopsy) within 4 weeks before first dose or planned during the trial
* Use of CYP3A4 strong inhibitor within 7 days or strong inducer within 21 days before first dose; use of anti-tumor Chinese medicine within 2 weeks before first dose or planned during the trial
* Participation in other clinical trials (investigational drug/device) within 4 weeks or 5 half-lives before first dose
* Use of other anti-tumor drugs within 14 days before first dose
* Spinal cord compression or symptomatic leptomeningeal metastasis
* Toxicity from previous anti-tumor therapy not recovered to ≤CTCAE Grade 1 (except alopecia or platinum-induced peripheral neuropathy)
* Symptomatic or unstable pleural/peritoneal effusion (stable ≥14 days after drainage is allowed)
* History of other malignancies (except cured malignancies with no recurrence in 5 years: cervical carcinoma in situ, basal cell carcinoma, papillary thyroid carcinoma)
* History of interstitial lung disease (ILD), drug-induced ILD, steroid-requiring radiation pneumonitis, or suspected ILD
* Uncontrolled severe systemic diseases (e.g., hypertension, diabetes, NYHA III-IV heart failure, unstable angina, myocardial infarction within 1 year, active bleeding)
* QTc >470 msec on resting ECG
* Clinically significant QT prolongation or arrhythmias increasing QT risk (e.g., complete left bundle branch block, III° AV block, congenital long QT syndrome, severe hypokalemia, use of drugs causing QT prolongation)
* Severe gastrointestinal dysfunction that impairs drug intake or absorption Infections requiring intravenous medication
* Active mental illness or drug addiction
* Known or suspected allergy to furmonertinib or its components
* Pregnant or lactating women; women or their partners planning pregnancy during the study
* Poor compliance (unable to follow study procedures)
* Other conditions deemed unsuitable for enrollment by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Median Progression-Free Survival (PFS) as assessed by Investigator | Approximately 18 months after the first patient begin study treatment
  The time from the first dose of the study drug to the progression of the disease (Investigator-Assessed) or death for any reason according to investigator.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) as assessed by RECIST 1.1 | Approximately 12 weeks following the first dose of study drug
  Proportion of subjects whose tumors were assessed as complete response(CR) or partial response(PR) according to RECIST 1.1.
Disease Control Rate (DCR) as assessed by RECIST 1.1 | Approximately 18 months from the first patient begin study treatment
  Proportion of subjects whose tumors were assessed as CR, PR or stable disease (SD) according to RECIST 1.1.
Central Nervous System (CNS) Objective Response Rate (CNS ORR) as assessed by RECIST 1.1 | Approximately 12 weeks after the first dose of study drug
  Proportion of subjects whose central nervous system (CNS) tumors (including intracranial parenchymal metastases and asymptomatic meningeal metastases as defined in the inclusion criteria) are assessed as Complete Response (CR) or Partial Response (PR) according to RECIST1.1.
Central Nervous System (CNS) Disease Control Rate (CNS DCR) as assessed by RECIST 1.1 | Approximately 18 months after the first dose of study drug
  Proportion of subjects whose central nervous system (CNS) tumors (including intracranial parenchymal metastases and asymptomatic meningeal metastases as defined in the inclusion criteria) are assessed as Complete Response (CR), Partial Response (PR), or Stable Disease (SD) according to RECIST 1.1.
Central Nervous System Progression-Free Survival (CNS PFS) as assessed by RECIST 1.1 | Approximately 18 months after the first dose of study drug
  The time from the first dose of the study drug (Furmonertinib) to the first occurrence of central nervous system (CNS) disease progression (assessed by RECIST 1.1) or death from any cause, whichever comes first.
Median Overall Survival (OS) | Approximately 24 months after the first dose of study drug
  The time from the first does of the study drugs to the death for any reason
Safety Profile (Adverse Events, AE) as assessed by CTCAE v5.0 | From the start of study drug to 28 days after the last dose of study drug
  The number of patients with adverse events and the severity grading (Grade 1-5) according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Progression Pattern as assessed by RECIST 1.1 and Clinical Evaluation | Approximately 18 months after the first dose of study drug
  Proportion of subjects with first disease progression classified as Intracranial, extracranial, or combined intracranial-extracranial progression.
Site Analysis of Disease Progression as assessed by RECIST 1.1 and Clinical Evaluation | Approximately 18 months after the first dose of study drug
  Frequency of specific progression sites.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) to be shared include demographic characteristics, clinical baseline data (e.g., ECOG PS score, EGFR mutation status, brain metastasis status), efficacy endpoints (median PFS, ORR, DCR, CNS ORR, CNS DCR, CNS PFS, OS) assessed by RECIST 1.1, adverse event data graded by CTCAE v5.0, progression pattern and site data, and biomarker (NGS) data collected at baseline and disease progression. The data will be made available after the completion of the primary analysis (expected by December 2028) for non-commercial scientific research purposes, to support further exploration of EGFR-mutated NSCLC with brain metastasis treatment.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Available from June 2029 (after completion of primary analysis) to December 2034 (5 years after data availability).
Access Criteria: Researchers interested in accessing the IPD must submit a formal research proposal to the leading research unit (Tianjin Medical University Cancer Institute and Hospital) and the sponsor for review. Approval will be granted based on the scientific merit of the proposal, alignment with the study's objectives, and compliance with data privacy and ethical requirements. A data use agreement (DUA) must be signed prior to data access, prohibiting re-identification of participants and restricting data use to non-commercial research.
URL: https://www.tjmuch.com/ipd-sharing-updates